CLINICAL TRIAL: NCT01256827
Title: Seven Year Observational Update of Macular Degeneration Patients Post-MARINA/ANCHOR and HORIZON Trials (SEVEN UP Study)
Brief Title: Seven Year Update of Macular Degeneration Patients
Acronym: SEVEN UP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IST-72116; FVF 4938s (Other: Genentech, Inc.)
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration; ranibizumab; geographic atrophy; ANCHOR Study; MARINA Study
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples will be drawn
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ranibizumab in MARINA/ANCHOR: Exudative AMD patients previously enrolled in the ranibizumab treatment arms of the MARINA or ANCHOR studies with subsequent enrollment into the HORIZON extension study.

SUMMARY:
The purpose is to assess long term vision outcomes and disease status in patients with age-related macular degeneration previously treated with ranibizumab as participants in the Phase 3 ANCHOR and MARINA Studies and the HORIZON Study.

DETAILED DESCRIPTION:
This is a cross-sectional cohort study of exudative age-related macular degeneration (AMD) patients seven or more years after initiation of the intravitreal ranibizumab regimen in the treatment arms of the pivotal ANCHOR or MARINA studies, who had subsequent follow up in the HORIZON Study. While the MARINA and ANCHOR studies established the benefit of ranibizumab at 2 years, many patients in the U.S. have now undergone treatment for many years, and the longer-term outcomes for this chronic disease remain unknown. Despite earlier hopes for limited duration treatment, subsequent clinical experience suggests that many patients require continued treatment. The patient population for this study is unique, in that the patients in the treatment arms of MARINA and ANCHOR are some of the earliest treated patients, providing the longest-term data available for AMD patients receiving ranibizumab. Patients recalled into this study will be evaluated to provide an update on their current visual acuity, disease activity status, anatomic characteristics, and genotype. There is a single study visit to extend the clinical history and to perform vision testing, ophthalmologic examination, and retinal imaging studies, including high-resolution spectral-domain OCT and fundus autofluorescence imaging, technologies unavailable at the time of the original ANCHOR and MARINA Trials. Genetic analysis will be performed for known AMD risk genes as well as candidate genes to study genotypic profiles associated with AMD disease progression and long-term treatment response. Understanding the course of 7-plus years of current generation AMD treatment will serve physicians in the ongoing management of this chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* previous participants in the ANCHOR or MARINA studies, and...
* who were assigned to one of the ranibizumab treatment arms, and...
* who were enrolled in the HORIZON extension study with a current SEVEN UP investigator
* ability to provide written informed consent and comply with study assessments

Exclusion Criteria:

* any separate ophthalmologic condition that the investigator believes would interfere with anatomic assessments in the trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exudative AMD patients who were previously participants in ranibizumab treatment arms of the ANCHOR or MARINA studies, and who subsequently enrolled in the HORIZON extension study
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
visual acuity 20/70 or better | at date of study visit
  percentage of study eyes with vision of 20/70 or better (ETDRS best-corrected vision with Snellen equivalent)

SECONDARY OUTCOMES:
mean change in visual acuity | at study visit
  Mean change in ETDRS best-corrected vision in study eyes, relative to baseline, exit from MARINA or ANCHOR, and exit from HORIZON
visual acuity 20/200 or worse | at date of study visit
  % of study eyes with ETDRS best-corrected visual acuity 20/200 or worse
visual acuity 20/40 or better | at date of study visit
  % of study eyes with ETDRS best-corrected visual acuity 20/40 or better
exudative AMD disease quiescence | at date of study visit and 6 months prior history
  % of eyes that have attained disease quiescence, defined by: 1) No leakage (SRF, PED, CME, CFT greater than 250 um on OCT) on clinical exam or on studies. 2) no subretinal intraretinal hemorrhage on clinical exam or FA, 3) Historical: none of the above in the last 6 months by chart review or history, and no treatment for exudative AMD within the last 6 months.
central geographic atrophy | date of study visit
  % of patients: 1) with central geographic atrophy (GA); 2) demonstrating progression of GA compared to baseline, exit from MARINA/ANCHOR, and exit from HORIZON; 3) with fellow eye GA development. GA measured by: fundus autofluorescence, high resolution OCT, and by interval comparison of fundus photography and fluorescein angiography
genotypic profile | date of study visit
  Genome-wide screening for high interest genes for associations with: geographic atrophy, disciform scar, current disease activity, therapeutic response to ranibizumab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Bhisitkul, MD, PhD, Principal Investigator — University of California, San Francisco; David S. Boyer, MD, Study Director — Retina-Vitreous Associates; SriniVas Sadda, MD, Study Director — USC Keck School of Medicine, Doheny Eye Institute; Kang Zhang, MD, PhD, Study Director — University of California San Diego, Shiley Eye Center
Locations (12):
- United States (12):
  - Retina-Vitreous Associates, Beverly Hills, California
  - USC Keck School of Medicine, Doheny Eye Institute, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - University of California San Francisco, San Francisco, California
  - Midwest Eye institute, Indianapolis, Indiana
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas